CLINICAL TRIAL: NCT01495962
Title: The Biomechanical Effects of Flaccid Paralysis Induced by Botulinum Toxin a After Damage Control Laparotomy: A Pilot Study
Brief Title: The Biomechanical Effects of Flaccid Paralysis Induced by Botulinum Toxin a After Damage Control Laparotomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Martin D. Zielinski, Assistant Professor of Surgery, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 10-008404
Record Dates: First submitted 2011-11-15; First posted 2011-12-20 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Wound; Abdomen, Abdominal Wall
Keywords: Damage Control Laparotomy; Open Abdomen; Botulinum Toxin A; Primary Fascial Closure
MeSH Terms: conditions — Wounds and Injuries | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botulinum Toxin A injection (Active Comparator)
  Interventions: Drug: Botulinum Toxin Type A
- Placebo (Normal Saline) injection (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Botulinum Toxin Type A — Six 25 cc injection of Botulinum Toxin A
  Arms: Botulinum Toxin A injection
Drug: Placebo — Placebo (Normal Saline)
  Arms: Placebo (Normal Saline) injection

SUMMARY:
Damage control laparotomy (DCL) is a life saving maneuver used with success in trauma and acute general surgery patients. The technique involves source control of sepsis and hemorrhage with an abbreviated laparotomy. In other words, the surgical procedure is cut short to allow for resuscitation in the ICU after the immediately life threatening pathology is treated. Planned re-exploration is then performed within 24-48 hours. It is at this procedure that the injuries are reconstructed. This technique, unfortunately, has several complications implicit with its use including wound infection, enterocutaneous fistula formation, and intra-abdominal abscess development.[1] Additionally, in patients whom primary fascial closure is not achieved, extensive abdominal wall reconstruction will be required in 6-12 months. The key for preventing these complications is definitive closure of the abdominal fascia, however, 10-50% of patients will have a planned ventral hernia with an open abdominal wound at dismissal [1,2] Proven methods for decreasing the rate of planned ventral hernia utilize tension in the midline to counter the effects of lateral abdominal muscular retraction.[3,4,5] Despite these improvements, however, the planned ventral hernia rate continues to be substantial.[2] Botulinum toxin a (BTX) is an FDA approved neuron modulating agent which has been used extensively in cosmetic, motor and pain disorders over the past 20 years [6,7]. The toxin blocks acetylcholine and pain modulator release (calcitonin gene related peptide and substance P) from the pre-synaptic cholinergic nerve terminal. The peptides are unable to bind at their motor end plate receptors through a process that cleaves proteins involved in the transport protein cascade. This results in flaccid paralysis and neuromodulation of the abdominal wall muscles resulting in reduced lateral tension and pain. Theoretically, this could increase the rates of primary fascial closure, improve pain sensation, decrease the rate of complications associated with open abdomens all while lowering the costs and need for future abdominal wall reconstruction.

ELIGIBILITY:
Inclusion Criteria

* male or female, aged ≥ 18 years or older
* signed Informed Consent form by appropriate patient representative
* undergone a DCL for trauma or acute general surgery

Exclusion Criteria

* death prior to BTX injection
* failure to achieve hemodynamic stability within 24 hours (stable or decreasing vasopressor support within 6 hours in combination with a stable or improving base deficit or lactate level)
* Viable pregnancy
* At risk populations (<18 years of age, prisoners)
* BMI > 50
* Pre-existing pareses (Amyotrophic Lateral Sclerosis, myopathies, motor polyneuropathies
* impaired neuromuscular transmission (Myasthenia Gravis, Lambert-Eaton Syndrome)
* concurrent aminoglycoside use
* chronic obstructive pulmonary disease
* known metastatic malignancy
* pre-existing cirrhosis
* necrotizing fasciitis of the trunk
* hypocoagulable state (INR >1.5)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to determine whether BTX will facilitate primary fascial closure after DCL. | 2 years
  The primary endpoint is the rate of delayed primary fascial closure. Delayed primary fascial closure will be considered when the rectus abdominus fascia is directly approximated in the midline during the same hospitalization as the initial DCL without the use of mesh.

SECONDARY OUTCOMES:
Non-invasive biomechanical testing results (surface wave elastography, traction index and durometry) | 2 years
Mortality | 2 years
Duration of mechanical ventilation | 2 years
Complications (wound infection, fascial dehiscence, enterocutaneous fistula formation, acute renal failure, pneumonia) | 2 years
Overall hospital cost | 2 years
Total narcotic use (morphine equivalents) | 2 years
ABPS score | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Martin D Zielinski, M.D., Principal Investigator — Mayo Clinic; David Dries, MD, Principal Investigator — Regions Hospital
Locations (2):
- United States (2):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Regions Hosptial, Saint Paul, Minnesota

REFERENCES:
- [Derived] Zielinski MD, Kuntz M, Zhang X, Zagar AE, Khasawneh MA, Zendejas B, Polites SF, Ferrara M, Harmsen WS, Ballman KS, Park MS, Schiller HJ, Dries D, Jenkins DH. Botulinum toxin A-induced paralysis of the lateral abdominal wall after damage-control laparotomy: A multi-institutional, prospective, randomized, placebo-controlled pilot study. J Trauma Acute Care Surg. 2016 Feb;80(2):237-42. doi: 10.1097/TA.0000000000000917. PMID 26813298